CLINICAL TRIAL: NCT01442350
Title: Myocardial Affectation in Patients With Fabry Disease Without Phenotypic Manifestation. Diagnostic Value of Biomarkers
Acronym: FAMY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Francisco Marín Ortuño (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other); Hospital General Universitario Elche (Other)
Responsible Party: Sponsor-Investigator, Francisco Marín Ortuño, Cardiologist, Hospital Universitario Virgen de la Arrixaca
Organization: Hospital Universitario Virgen de la Arrixaca (Other)
Other Study IDs: Fabry-Myocardial
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Fabry Disease, Cardiac Variant; Right Ventricular Hypertrophy
Keywords: Fabry disease; annexin 5; miosin; sarcoma; alfa-galactosidase; fibrosis; apoptosis; biomarkers; NT-proBNP
MeSH Terms: conditions — Fabry Disease, Cardiac Variant; Hypertrophy, Right Ventricular; Fabry Disease; Sarcoma; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genotyping of relatives of mutation-known Fabry probands: in order to know which are the relatives carrying mutations. (The investigators have already started this task).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The cardiac variant of the Fabry disease is a rare cardiomyopathy affecting 1/50000 individuals in general population. It is generally diagnosed in advanced stages of the disease, because it presents clinical features very similar to the hypertrophic cardiomyopathy ones, making difficult the correct diagnosis. In Fabry disease there is a remodeling process of the myocardial interstitium and apoptosis of myocytes which leads to fibrosis development and later systolic dysfunction. The investigators propose to evaluate the utility of several biomarkers in the diagnosis of this cardiomyopathy, to facilitate the early diagnosis, which is clue to establish early enzyme replacement therapy or intensify the patients' follow up. In order to achieve this objective, the investigators will analyze markers of endothelial dysfunction, fibrosis and apoptosis in peripheral blood samples of patients carrying the mutation but without clinical manifestations and the investigators will compare their levels with dose obtained from two different control groups: diagnosed patients presenting clinical manifestations or index cases and healthy controls without carrying the mutation.

DETAILED DESCRIPTION:
Fabry disease is an X-linked recessive disease, affecting lysosomal storage with a variable phenotype characterized by the accumulation of glycosphingolipids in several tissues. It has been described more than 200 mutations in the alfa-galactosidase A (GLA) gene which cause Fabry disease. Nowadays, the treatment of Fabry disease consists of enzyme replacement therapy (ERT) which development has shown a reversal of abnormal accumulation of glycosphingolipids in different tissues and a clinical improvement or stabilization (1). Unlike classic systemic Fabry disease with multiple organ affectation, the cardiac variant of the disease is characterized by myocardial hypertrophy. Hence, cardiac Fabry variant is defined as a storage myocyte disorder mimicking the clinical features of the hypertrophic cardiomyopathy (HCM)(2).

The gold standard for the diagnosis of Fabry disease is the electron microscopy evaluation of cardiac samples obtained from endomyocardial biopsy (2), although it has been published that the determination of the alfa-galactosidase activity in plasma of patients diagnosed of Fabry disease, followed by sequencing of the GLA gene in those individuals with low activity level is a good non-invasive diagnostic method which allows the identification of the disease carriers and the early start of the enzymatic replacement therapy (3).

Due to the similarity between clinical characteristics of both diseases and to the extraordinary low incidence of the Fabry disease, the biopsy execution is rarely carried out for diagnosis. Hence, it has been speculated that a higher disease incidence should exist hidden among patients presenting with clinical symptoms of HCM. Several studies have evaluated the incidence of the Fabry disease among patients diagnosed of HCM, finding out that even 8-10% of these patients actually presented Fabry disease (4,5), although a bias in the patient selection can exist. In more recent studies including one carried out by our group with a higher number of patients, a lower incidence (between 1-3%) has been found (3,6). So, Fabry is a rare disease affecting 1/50000 individuals in the population (3).

Extracellular matrix is a dynamic structure with an intense participation in the myocardial remodeling that occurs in different cardiovascular diseases (7). Alterations in the extracellular matrix could perform an important role in the diastolic dysfunction process linked to the myocardial hypertrophy. Collagen deposits increase left ventricular chamber stiffness and ventricular load during diastole is compromised. Collagen turnover is increased when compared to healthy controls, and synthesis is predominant over degradation, finding associated changes in metalloproteinase activity (MMP, which are the principal enzymes in charge of matrix degradation) and their inhibitors (TIMP) (8). Our group has recently published several papers about the relevance of the fibrosis in patients with MCH (9,10,11,12). The investigators found out that fibrosis, assessed by late Gadolinium enhancement in cardiac magnetic resonance, is related to ventricular remodeling, hypertrophy, ventricular tachycardia (10) and functional state of the patient (11) and that MMP-9 value is independently associated to fibrosis (9). There are also studies describing structural changes in the matrix associated to Fabry disease, where fibrosis presence is evident both at the interstitial level and replacing myocardiocytes loss (13). However, it has not been yet demonstrated whether the alteration in the interstitial matrix takes place due only to fibroblasts activation in response to humoral or mechanical factors without myocardiocytes loss or, on the contrary, it is associated to cellular death.

The interest of apoptosis, or programmed cell death, is increasing in heart failure. Apoptosis can be activated by the interaction of cell surface death receptors (i.e. receptors of tumoral necrosis factor superfamily -TNFR- and Fas protein receptor), with its ligands (TNF-alfa and Fas ligand, FasL) (14), and by activation of the mitochondrial pro-apoptotic mechanisms, in response to unfavorable changes in intracellular environment (15). The subsequent development is regulated by the Bcl-2 protein group (16) and executed by the caspase family (17). During the apoptosis, Annexin 5, is produced in the myocytes and secreted to the interstitial space (18,19). Annexin 5 seems to contribute to the intracellular calcium management alteration, leading to the systolic dysfunction (20, 21). Myocardiocytes death via apoptosis could be a more common process that previously thought, with estimation of repair process that contribute to the interstitium expansion. GDF-15 is a member of the TGF-β superfamily, and a well establish marker of risk and prognosis in acute coronary syndromes. It has been recently proposed as a regulator of fibrosis and tissue remodeling processes probably by prevention of apoptosis (22). Apoptosis of myocardiocytes leads to the progressive ventricular wall slimming, as previously reported in MCH (23), and systolic dysfunction.

Many of the molecules involved in apoptosis and ventricular remodeling can be detected in peripheral blood and are known as biomarkers. Biomarkers give information about normal biological processes or physiopathologic mechanisms and can be very useful in differential diagnosis or even in prognosis. Nowadays, there is a raising interest in the study and utility of biomarkers in cardiovascular disease, being more used in ischemic cardiopathy and heart failure (24-27). Unfortunately their study in HCM has been less developed, even less in Fabry disease. Brain natriuretic peptide (BNP) is the most studied biomarker in HCM and has been related to the presence of heart failure symptoms (28-30), poor functional capacity (30) and left ventricular outflow obstruction (31-34). On the other hand ST2 has started very recently to be considered as a good biomarker for myocardial-specific response to stretch, with synergistic implications in prognosis with BNP (35).

Our group is currently developing a project studying several biomarkers (myocardial stress, endothelial damage, hypercoagulable state) in order to explore different systems involved in ventricular remodeling in HCM (assessed by echocardiography and cardiac magnetic resonance) that could be very similar in Fabry disease.

In Fabry disease, plasma or urine level of globotriaosylceramide (Gb3) is used as biomarker. This glycosphingolipid is stored in lysosomes in Fabry patients, although is has been shown that detected plasma or urine concentrations can vary, due to different mutations that do not provoke a complete loss of alfa-galactosidase activity. In addition, in heterozygous women plasma levels can be normal but there are some data suggesting high concentration in urine (36). On the other hand, it has been suggested that is lactosylceramide, a catabolic product of Gb3, who regulates the expression pattern of TNF-alfa and y ICAM-1, contributing to atherosclerosis development (37).

The investigators dispose of a specialized cardiomyopathy clinic in each of the three hospitals: Hospital Universitario Virgen de la Arrixaca, Murcia, Hospital General Universitario de Alicante, and Hospital General Universitario de Elche. The investigators have already recruited 12 families with diagnosed Fabry probands and a total of 60 relatives clinically checked up within last 4 months. The investigators consider that the recruitment of patients has been successful and are ready to carry out the present project. However, the investigators would like to participate with other centres in order to share patients and mutated relatives without phenotypic disease expression.

The aim of the present project is to study biomarkers of apoptosis, fibrosis and interstitial remodeling in peripheral samples of patients diagnosed with Fabry disease and relatives. Our objective is to establish whether exists or not myocardial affectation data in mutations carriers without phenotypic disease criteria. The investigators will also focus on different polymorphisms and their implication in the development of Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* 20 families with Fabry diagnosed probands, including up to 80 relatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This task will be performed at the monographic hypertrophic cardiomyopathy clinic. The investigators intention is to include 12 families for testing the biomarkers elevation correlation with the presence of disease. The investigators plan to achive the inclusion of 30 families with Fabry diagnosed probands, including up to 130 relatives for verification and the polimorfisms' study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)